CLINICAL TRIAL: NCT05059249
Title: Effects of Mechanical Versus Manual Traction in the Management of Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2021/5
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical; Disc Degeneration; Disc Prolapse; Disc Prolapse With Radiculopathy; Lumbar Radiculopathy
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Radiculopathy | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Traction (Experimental): Moist heat packs & TENS for ten minutes followed by Manual Traction and 3 sets of slow gentle segmental mobilizations (unilateral and posterior-anterior) with at least 10 to 15 repetitions firstly but modified as per the response of the patient.
  Interventions: Procedure: Hot Pack; Procedure: Manual Traction; Procedure: Joint Mobilization; Procedure: TENS
- Mechanical traction (Experimental): Moist heat packs & TENS for ten minutes followed by Mechanical Traction and 3 sets of slow gentle segmental mobilizations (unilateral and posterior-anterior) with at least 10 to 15 repetitions firstly but modified as per the response of the patient
  Interventions: Procedure: Hot Pack; Procedure: Mechanical Traction; Procedure: Joint Mobilization; Procedure: TENS

INTERVENTIONS:
Procedure: Hot Pack — Superficial Heating
Procedure: Manual Traction — Manual Traction for 10 minutes
  Arms: Manual Traction
Procedure: Mechanical Traction — Mechanical Traction for 10 minutes
  Arms: Mechanical traction
Procedure: Joint Mobilization — 3 sets of slow gentle segmental mobilizations (unilateral and posterior-anterior) with at least 10 to 15 repetitions
Procedure: TENS — TENS for 10 minutes with hot pack

SUMMARY:
This study compared the effects of mechanical and manual traction on pain, disability and lumbar spinal curvature in patients with discogenic low back pain

ELIGIBILITY:
Inclusion Criteria:

* Patients with discogenic low back pain,
* Patients of both genders
* Age ranges from 20 to 60 years
* NPRS > 5

Exclusion Criteria:

* Patients with non-mechanical back pain
* Patients with known metabolic diseases,
* Osteoporotic patients,
* Recent history of spinal trauma or surgery,
* Lumbar myelopathy,
* Cauda equine syndrome.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. Where 0 indicate no pain and 10 indicate severe pain.
Oswestry disability index | 6 weeks
  Changes from base line The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Furqan Yaqoob, PhD*, Principal Investigator — Foundation University Islamabad; Muhammad Osama, PhD*, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No